CLINICAL TRIAL: NCT03615300
Title: Predicting Long-term Outcomes After Cardiac Arrest by Using Serum NGAL: A Prospective, Observational Study
Brief Title: Predicting Long-term Outcomes After Cardiac Arrest by Using Serum NGAL
Status: Terminated | Type: Observational
Why Stopped: Recruiting unavailable
Sponsor: Uijeongbu St. Mary Hospital (Other)
Responsible Party: Principal Investigator, Joo Suk Oh, MD. PhD., Professor, Uijeongbu St. Mary Hospital
Other Study IDs: UC18OESI0055
Record Dates: First submitted 2018-07-30; First posted 2018-08-03 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Out-of-Hospital Cardiac Arrest
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- good neurologic outcome: Patients with good neurological prognosis after 6 months (CPC 1, 2). serum NGAL is collected.
  Interventions: Diagnostic Test: serum NGAL
- poor neurologic outcome: Patients with poor neurological prognosis after 6 months (CPC 3, 4, 5). serum NGAL is collected.
  Interventions: Diagnostic Test: serum NGAL

INTERVENTIONS:
Diagnostic Test: serum NGAL — serum NGAL was measured at 0, 24, 48, and 72 hours after recovery of spontaneous circulation.

SUMMARY:
This study was performed to determine the prognosis of patients after cardiac arrest using serum markers called NGAL. The initial NGAL values of patients with post-cardiac arrest syndrome are checked by blood tests, and the long-term neurological prognosis and survival rate are collected after 6 months.

DETAILED DESCRIPTION:
Serum NGAL is currently being used as a test to determine the likelihood of developing renal failure. However, in a previous study, serum NGAL correlated with neurological prognosis in post cardiac arrest syndrome patients. This prospective study attempts to see the role of serum NGAL as a prognostic factor by including a sufficient number of patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who underwent targeted temperature management after out-of-hospital cardiac arrest.

Exclusion Criteria:

* Patients who did not survived 3 days after cardiac arrest.
* Pre-existing end-stage renal disease or dependence on renal replacement therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult survivors after out-of-hopital cardiac arrest who underwent targeted temperature management and survived longer than 3 days.
Sampling Method: Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2018-06-28 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Long term neurologic outcome | 6 months
  Patients' CPC score after 6 months (good outcome : CPC score 1, 2 / poor outcome : CPC score 3, 4, 5)

SECONDARY OUTCOMES:
Proportion of participants with Overall Survival at 6 months | 6 months
  6-month survival rate of patients'

CONTACTS AND LOCATIONS:
Overall Officials: Joo Suk Oh, MD PhD, Principal Investigator — The Catholic University of Korea, Uijeongbu ST. Mary's Hospital
Locations (1):
- Uijeongbu St. Mary's Hospital, Uijeongbu-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Elmer J, Jeong K, Abebe KZ, Guyette FX, Murugan R, Callaway CW, Rittenberger JC; Pittsburgh Post-Cardiac Arrest Service. Serum Neutrophil Gelatinase-Associated Lipocalin Predicts Survival After Resuscitation From Cardiac Arrest. Crit Care Med. 2016 Jan;44(1):111-9. doi: 10.1097/CCM.0000000000001357. PMID 26457752
- [Result] Park YR, Oh JS, Jeong H, Park J, Oh YM, Choi S, Choi KH. Predicting long-term outcomes after cardiac arrest by using serum neutrophil gelatinase-associated lipocalin. Am J Emerg Med. 2018 Apr;36(4):660-664. doi: 10.1016/j.ajem.2017.12.013. Epub 2017 Dec 7. PMID 29317152